CLINICAL TRIAL: NCT00014456
Title: A Dose-Escalation Trial Of The Combination Of Docetaxel, Gemcitabine And Filgrastim (NEUPOGEN) For The Treatment Of Patients With Advanced Solid Tumors
Brief Title: Combination Chemotherapy Plus Filgrastim in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9933; P30CA023108 (NIH); DMS-9933; NCI-G01-1933
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Bladder Cancer; Breast Cancer; Carcinoma of Unknown Primary; Esophageal Cancer; Gastric Cancer; Head and Neck Cancer; Lung Cancer; Melanoma (Skin); Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Sarcoma
Keywords: stage IV breast cancer; recurrent breast cancer; stage IV gastric cancer; recurrent gastric cancer; metastatic osteosarcoma; recurrent non-small cell lung cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; chondrosarcoma; recurrent adult soft tissue sarcoma; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; recurrent osteosarcoma; recurrent bladder cancer; stage IV bladder cancer; stage IV prostate cancer; recurrent prostate cancer; stage IV melanoma; recurrent melanoma; stage IV non-small cell lung cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; classic Kaposi sarcoma; AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma; recurrent metastatic squamous neck cancer with occult primary; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; stage IV uterine sarcoma; recurrent uterine sarcoma; borderline ovarian surface epithelial-stromal tumor; recurrent carcinoma of unknown primary; ovarian sarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; recurrent mucoepidermoid carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV adult soft tissue sarcoma; stage IV pancreatic cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Neoplasms, Unknown Primary; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Melanoma; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Sarcoma; Osteosarcoma; Carcinoma, Non-Small-Cell Lung; Chondrosarcoma; Carcinoma, Ovarian Epithelial; Small Cell Lung Carcinoma; Salivary Gland Neoplasms; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi; Neuroectodermal Tumors, Primitive, Peripheral; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory | interventions — Filgrastim; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy plus filgrastim in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of docetaxel in combination with gemcitabine and filgrastim (G-CSF) in patients with advanced solid tumors.
* Determine the dose-limiting toxicity associated with this regimen in these patients.
* Assess the objective anti-tumor response in patients treated with this regimen.
* Determine fatigue and blood cytokines in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of docetaxel.

Patients receive docetaxel IV over 1 hour followed by gemcitabine IV over 30 minutes on day 1. Patients also receive filgrastim (G-CSF) subcutaneously daily beginning on day 2 and continuing until blood counts recover. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Fatigue is assessed at baseline and then at weeks 2, 5, 7, and 9 during therapy.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study within 15-22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor that is not curable by surgery or radiotherapy

  * Sarcoma
  * Melanoma
  * Carcinoma of unknown primary
  * Pancreatic cancer
  * Lung cancer
  * Ovarian cancer
  * Breast cancer
  * Bladder cancer
  * Gastric cancer
  * Esophageal cancer
  * Prostate cancer
  * Head and neck cancer
* No hematopoietic or lymphoid tumors
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 60-100%
* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST and/or ALT no greater than 5 times upper limit of normal (ULN) if alkaline phosphatase no greater than ULN OR
* Alkaline phosphatase no greater than 5 times ULN if AST and ALT no greater than ULN OR
* AST and/or ALT no greater than 1.5 times ULN if alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 2 times ULN OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No congestive heart failure
* No unstable angina

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No known sensitivity to E. coli-derived products

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 2 weeks since prior cytotoxic anti-tumor therapy (4 weeks for nitrosourea or mitomycin) and recovered
* No prior docetaxel or gemcitabine

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Determine the maximal tolerated dose of docetaxel in combination with gemcitabine given intravenously every 2 weeks with pegfilgrastim support | Four years
Define dose limiting adverse events associated with the combination | Four years

SECONDARY OUTCOMES:
Objective antitumor response | Four years

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin H. Dragnev, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Dragnev KH, Hardin SB, Pipas JM, Davis TH, Rigas JR. A dose escalation trial of biweekly docetaxel and gemcitabine with filgrastim or pegfilgrastim for the treatment of patients with advanced solid tumors. Chemotherapy. 2010;56(2):135-41. doi: 10.1159/000313526. Epub 2010 Apr 20. PMID 20407240